CLINICAL TRIAL: NCT01630343
Title: The Efficacy of Pain Management Protocol for Elderly Hip Fracture Patients After Surgery: A Prospective Cohort Study
Brief Title: Pain Management in Geriatric Hip Fracture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Elizabeth Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Ho Chin Hung, Associate Consultant (Orthopaedics and Traumatology), Queen Elizabeth Hospital, Hong Kong
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QEHHIPPAIN
Record Dates: First submitted 2012-06-20; First posted 2012-06-28 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Geriatric Hip Fracture Pain Management
Keywords: Geriatric hip fracture; pain management
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; Tramadol; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regular oral Panadol and Tramadol (Experimental): Geriatric (age >65) Patient having traumatic hip fracture will have three weeks of regular prescription of oral Panadol(500mg) and tramadol (50mg) three times a day. Operation will be done within 3 days usually followed by rehabilitation period.
  Interventions: Drug: Panadol 500mg tablet, tramadol 50mg capsule
- Panadol and tramadol oral in prn basis (Experimental): Control group is that patient having geriatric hip fracture will have oral analgesics ( Panadol 500mg Q4H and tramadol 50mg Q4H ) in prn basis.
  Interventions: Drug: Paracetamol tablet and Tramadol capsule

INTERVENTIONS:
Drug: Paracetamol tablet and Tramadol capsule — Panadol 500mg tablet Q4H prn Tramadol 50mg capsule Q4H prn
  Other Names: Endpain, tramadol
  Arms: Panadol and tramadol oral in prn basis
Drug: Panadol 500mg tablet, tramadol 50mg capsule — Regular Panadol 500mg tds with tramadol 50mg capsule tds for 3 weeks after injury
  Other Names: Endopain, tramadol
  Arms: Regular oral Panadol and Tramadol

SUMMARY:
The Null Hypothesis is that there is no association between Pain regime and the functional performance among geriatric patients having traumatic hip fracture. Two limbs are being assessed:1. Three weeks of regular oral Panadol and Tramadol after hip fracture 2. Oral Panadol and tramadol taking in p.r.n. basis. Functional outcome including Numerical Rate Scale for pain assessment, Functional Independency Measure and Elderly Mobility Score are chosen.

DETAILED DESCRIPTION:
200X2 patients are recruited during two periods within the study period where regular oral analgesics is given for the first 200 patients while the rest of patient will receive oral analgesics upon demand

ELIGIBILITY:
Inclusion Criteria:

* Both sex of Age > 65
* Traumatic non-pathological fracture neck of femur or trochanteric or subtrochanteric fracture having operative intervention

Exclusion Criteria:

* Age < 65
* Pathological fracture
* Multiple lower limb fractures
* Old fracture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Functional Independency Measure(FIM) | 2 years
  FIM including motor and cognitive function of a patient. Motor area covers self care, ambulation, bowel and bladder and etc.
Elderly Mobility Score | 2 years
  It is to assess mobility in frail elderly people. A final score rangeing from 0-20 is assigned during several time-point of rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Chin Ping Hong, Raymond, FRCSE(Edin), Study Director — The Queen Elizabeth Hospital
Locations (1):
- Department of Orthopaedics and Traumatology, Queen Elizabeth Hospital, Hong Kong SAR, China